CLINICAL TRIAL: NCT01089491
Title: Localization and Characterization of Cells in the Lumbar Epidural Cavity of Patients With Low Back Pain With or Without Radiculopathy
Brief Title: Study of Cells From Spinal Cavity of Patients With Low Back Pain
Status: Withdrawn | Type: Observational
Why Stopped: PI chose not to conduct the study; no data collected.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: James Heavner, DVM, PhD/Professor, Director of Research, Texas Tech University Health Sciences Center
Other Study IDs: L10-081
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Epiduroscopy; Cytology; Electrical stimulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Up to two (2) cell samples will be collected from different sites in the epidural space
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study to determine if cells collected give us information about what is causing a patient pain can be detected and connected with epiduroscopy images (pictures taken with a small fiber optic scope). We want to determine if abnormal areas are the source of that pain by using a catheter to provide a brief, low intensity electrical stimulation. We also want to determine if there are cells in the epidural cavity (area surrounding the spinal cord) of patients who have low back pain with or without pain shooting down one or both legs that provide information about what is causing the pain.

DETAILED DESCRIPTION:
The pain group at TTUSOM has pioneered a treatment for low back pain with or without radiculopathy called epidural neurolysis (or other names, e.g.: lysis of epidural adhesions, the Racz procedure). This technique is now used worldwide. The treatment is based on substantial evidence that pathological processes within the epidural space innate and sustain pain. The goal of epidural neurolysis is to deposit therapeutic agents directly into the area of pathology (i.e., targeted drug delivery). The procedure involves documentation via epidurograms that radio opaque material injected into the epidural space prior to treatment does not enter the suspected area of pathology. This area is determined by signs and symptoms revealed by the patient history and physical examination.

After a filling defect that corresponds to the suspected area of pathology is documented by epidurography, a specially designed catheter is directed into the defect. Mechanical forces applied by the catheter and hydraulic forces applied by injection of isotonic saline through the catheter as well as injection of hyaluronidase, are used to enter and remove barriers to targeted delivery of drug. Next drugs, usually corticosteroid, local anesthetic and hypertonic saline, are injected to treat what is presumed to be inflammation and edema.

More recently, epiduroscopy has been introduced as an aid to epidural neurolysis. Epiduroscopy allows visual inspection of epidural tissue. Epiduroscopy is performed by inserting a flexible endoscope through the sacral hiatus. Using epiduroscopy, we and others have observed change in the epidural space that we believe are related to the etiology of the pain. We see changes consistent with various stages of inflammation either acute or chronic. We see increases in vascularity, displacement of fat by fibrous tissue as well as changes in the texture and color of peridural fat.

We have developed a method for retrieving cells from suspected areas of pathology and of culturing the cells via the working channel of the epiduroscope using a cytology brush. The collected cells are characterized to establish a diagnosis and to aid treatment.

To confirm areas which appear to be abnormal when viewed via epiduroscopy are involved in the painful condition for which the patient is seeking treatment, we test the area with hydrostatic pressure (saline injection) or by touching with the epiduroscope tip (mechanical stimulation). These stimuli do not normally elicit pain. However, when the stimulus does elicit pain in the region of the painful region of the patient's body, the abnormal appearing tissue in the epidural space is considered to be involved in painful process affecting the patient. This is similar to "pain mapping" done by others when electrical stimulation is used to search for the area of pathology. Adapting this approach, applying electrical stimulation via a stimulating probe (FDA approved) inserted through the working channel of the epiduroscope will allow more precise localization of pathological tissue than does the methods we currently use.

We will collect cells during epiduroscopy and characterize them in vitro. A new dimension of this project is to deliver electrical stimulation to more accurately locate the source of pain from where cells should be sampled.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent and HIPAA forms
* Age >18 years at the time of signing the informed consent
* Scheduled for epiduroscopy assisted epidural neurolysis
* A diagnosis of low back pain with or without radiculopathy

Exclusion Criteria:

* Not scheduled for epiduroscopy assisted epidural neurolysis
* In the opinion of the investigator, the patient's overall condition is not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients receiving outpatient lysis of adhesions treatment at University Medical Center in Lubbock TX.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Characteristics of cell types | 6 months
  We expect that cell types identified will vary some from patient to patient depending in part upon how acute or chronic is the patient's disease and whether or not the patient has had prior surgery. We expect the cells will indicate that a pathological process is present and will provide information about the characteristics of the process.

SECONDARY OUTCOMES:
Electrical stimulation to locate pain | 6 months to 1 year
  We expect that electrical stimulation will improve the precision with which abnormal, painful structures are localized and thereby improve collection of cells directly involved in the patient's pain.

CONTACTS AND LOCATIONS:
Overall Officials: James E Heavner, DVM, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States